CLINICAL TRIAL: NCT05229471
Title: Management of Recurrent Venous Thromboembolism During Anticoagulant Treatment in Cancer Patients - a Prospective Cohort Study
Acronym: REDUCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Harry R. Buller, Professor of Internal Medicine, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W19_237
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cancer; Venous Thromboembolism; Recurrence
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: To prospectively evaluate clinical outcomes during guideline-recommended LMWH dose escalation for recurrent VTE during LMWH or DOAC treatment for cancer-associated thrombosis.

Study design: International, prospective, observational cohort study Study population: Adult cancer patients with symptomatic or incidental recurrent VTE while receiving LMWH or DOACs for acute VTE are eligible. Main exclusion criteria include anticoagulant treatment for the recurrent VTE for more than 72 hours, severe hepatic dysfunction, active bleeding, recent major surgery, uncontrolled hypertension, known bleeding diathesis, and a life expectancy of less than 1 month.

Study procedures: Patients will be managed at the discretion of the treating physician, who will be encouraged to follow guideline recommendations. These guidelines suggest supra-therapeutic dose LMWH for 4 weeks (+/- 5 days) followed by therapeutic dose LMWH or therapeutic dose DOAC, while it is suggested to treat patients with VTE recurrence during maintenance dose LMWH (i.e. 75 to 80% of full therapeutic weight adjusted dose) with therapeutic dose of LMWH or DOAC.

Main study parameters/endpoints: The co-primary outcomes are new symptomatic or incidental recurrent VTE during 3 months of follow-up and on-treatment major bleeding. Secondary outcomes include recurrent incidental VTE, recurrent symptomatic VTE, recurrent incidental or symptomatic proximal or distal DVT, recurrent incidental or symptomatic PE, clinically relevant non-major bleeding, all-cause mortality, and cancer-related mortality. VTE occurring at other sites such as cerebral DVT or splanchnic DVT will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Documented active cancer (i.e. diagnosis of cancer within the past 6 months; recurrent, regionally advanced, or metastatic disease; currently receiving treatment or received treatment within the past 6 months)
* Objectively confirmed symptomatic or incidental recurrent VTE while on anticoagulant therapy. The previous VTE and index recurrent VTE will include symptomatic or incidentally detected proximal deep vein thrombosis (DVT) of the lower extremities; symptomatic proximal upper extremity DVT (either related to a catheter or not); symptomatic distal DVT; symptomatic or incidentally detected multiple subsegmental, segmental or more proximal pulmonary embolism (PE).

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Use of thrombolysis
* Anticoagulant treatment for the recurrent VTE for longer than 72 hours
* Treatment with fondaparinux, unfractionated heparin, prophylactic doses of LMWH, or VKAs at time of recurrent VTE
* Acute hepatitis, chronic active hepatitis, or severe hepatic dysfunction (Child Pugh C or <MELD > 10)
* Active bleeding
* Recent major surgery (<2 weeks or longer, if still at high risk for bleeding)
* Uncontrolled hypertension (systolic arterial pressure >160 mmHg)
* Known bleeding diathesis
* Platelet count <50.000 mm3
* Creatinine clearance <30 mL/min (Cockcroft-Gault formula)
* Life expectancy of less than 1 month
* Dual antiplatelet therapy or aspirin at doses ≥165 mg daily
* Current diagnosis or history of heparin-induced thrombocytopenia
* Any condition, which in the opinion of the investigator, would put the subject at an unacceptable risk from participating in the study.
* Suspected non-compliance at the time of recurrent VTE

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected adult cancer patients who develop symptomatic or incidental recurrent VTE while receiving appropriate doses of LMWH or DOACs for an acute VTE.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent venous thromboembolism | 90 days
  objectively confirmed recurrent VTE
Major bleeding | 90 days
  Major bleeding per ISTH criteria

SECONDARY OUTCOMES:
Clinically relevant non-major bleeding | 90 days
  CRNMB per ISTH criteria

CONTACTS AND LOCATIONS:
Locations (9):
- Gabriele D'Annunzio University, Chieti, Italy
- Netherlands (3):
  - Meander Medisch Centrum, Amersfoort
  - Amsterdam UMC, location AMC, Amsterdam
  - Leids Universitair Merisch Centrum, Leiden
- Spain (5):
  - Hospital Universitario Puerto Real, Cadiz
  - hospital general universitario de Elche, Elche
  - Clínica Universidad Navarra en Madrid, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Undecided
Researchers are open to discussing plans for data sharing on IPD analysis.